CLINICAL TRIAL: NCT06199583
Title: Diagnostic Value of Shear-Wave Elastography for Patellar Tendinopathy in Female Volleyball and Basketball Athletes
Brief Title: Diagnostic Value of Shear-Wave Elastography for Patellar Tendinopathy
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sergen Devran, Sports Medicine Specialist, Istanbul University
Other Study IDs: IstanbulU-SportsMedicine
Record Dates: First submitted 2023-12-17; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Patellar Tendinopathy
Keywords: Patellar tendinopathy; shear-wave elastography; ultrasound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patellar tendinopathy: Contains athletes with patellar tendinopathy
  Interventions: Diagnostic Test: Shear-wave elastography
- Non-patellar tendinopathy: Contains athletes without patellar tendinopathy
  Interventions: Diagnostic Test: Shear-wave elastography

INTERVENTIONS:
Diagnostic Test: Shear-wave elastography — Ultrasound shear-wave elastography

SUMMARY:
To investigate the accuracy of shear-wave elastography (SWE) in diagnosing patellar tendinopathy in female volleyball and basketball players. In addition, we want to compare different parts of the patellar tendon and investigated the effects of different knee angles.

ELIGIBILITY:
Inclusion Criteria were:

* being a female athlete between the ages of 17-35 playing professional basketball or volleyball and agreeing to participate in the study

Exclusion Criteria were:

* to have a history of partial or full-thickness patellar tendon tear,
* if they received an injection in or around the patellar tendon within the past 12 months,
* undergone patellar tendon graft repair for anterior cruciate ligament, had a ligament or meniscus operation within the past six months,
* have a chronic disease (such as diabetes, heart disease, or rheumatic disease),
* are actively using oral contraceptives,
* have an active infection in the knee or surrounding tissues

Ages: 17 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: female athletes between the ages of 17-35 playing professional basketball or volleyball.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Shear-wave elastography | Through study completion, an average of 3 months
  Ultrasound shear-wave elastography
Ultrasound | Through study completion, an average of 3 months
  Tendon thickness, hypoechoic region, power doppler

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Faculty of Medicine Sports Medicine Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No